CLINICAL TRIAL: NCT06456203
Title: Artificial Intelligence for Chest Radiography: Impact on Economics, Patient Outcomes and Radiology Service Delivery
Brief Title: Trial of Artificial Intelligence for Chest Radiography
Acronym: ACER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Charlene Liew, Clinical Assistant Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023/2280
Record Dates: First submitted 2024-06-04; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Pneumonia; Lung Cancer
Keywords: Radiology; artificial intelligence; triage; radiography
MeSH Terms: conditions — Pneumonia; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (No Intervention): Chest radiographs reported with AI assistance
- AI assisted (Active Comparator): AI assisted detection, triage and reporting of CXR
  Interventions: Diagnostic Test: AI

INTERVENTIONS:
Diagnostic Test: AI — Artificial intelligence triage and reporting system
  Arms: AI assisted

SUMMARY:
Randomized Clinical Trial of the impact of Chest radiograph AI-assisted triage and report generation upon clinical outcomes and an economic analysis of impact of AI decision support on radiology service delivery.

DETAILED DESCRIPTION:
Randomized, prospective selection of patients. Control group involves radiologists reporting chest radiographs as per reference standard clinical workflow Intervention group involves radiologists assisted with AI reporting an AI-triaged worklist of chest radiographs using an AI report generation tool Clinical outcomes on patients are studied at pre-determined study endpoints, including time to discharge from the hospital and re-admission rates.

Economic analysis on cost-avoidance from man-hours saved from report generation and triage.

ELIGIBILITY:
Inclusion Criteria:

* All patients attending radiography to have chest radiographs during the study period

Exclusion Criteria:

* age below 14
* deceased before discharge
* chest radiograph performed in non-standard projections

Ages: 14 Years to 130 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Report generation time | 12 months
  Time for radiologist to produce each individual CXR report
Turnaround Time | 12 months
  Time from patient arrival at radiography department to time for clinical team to receive report
Time to discharge | 12 months
  Time from patient arrival at radiography department to time to discharge from hospital

SECONDARY OUTCOMES:
30-day patient readmission rate | 12 months
  Rate of readmission of patient to hospital after discharge within 30 days

IPD SHARING:
Plan to Share IPD: No